CLINICAL TRIAL: NCT00823485
Title: Clinical Efficacy of In-situ Thrombolysis in Case of Intraventricular Haemorraghia by Aneurysm Rupture
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 05-CIR-03
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Aneurysm, Ruptured; Subarachnoid Hemorrhage
MeSH Terms: conditions — Aneurysm, Ruptured; Subarachnoid Hemorrhage | interventions — Fibrinolysis; Drainage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): drainage of hemorraghia
  Interventions: Procedure: drainage
- 1 (Experimental): Actylise
  Interventions: Procedure: fibrinolysis in situ

INTERVENTIONS:
Procedure: fibrinolysis in situ — intraventricular injection of actilyse
  Arms: 1
Procedure: drainage — drainage
  Arms: 2

SUMMARY:
The purpose of this study is to determine the impact of in situ fibrinolysis on the mortality at 30 days in case of subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* subarachnoid hemorrhage by aneurysm rupture
* severe intraventricular hemorraghia

Exclusion Criteria:

* pregnant women
* hemostasis disturbance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
assessment of mortality | at 30 days

SECONDARY OUTCOMES:
assessment of morbidity | at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Neurosurgery department , Nice University Hospital, Nice, France

REFERENCES:
- [Derived] Litrico S, Almairac F, Gaberel T, Ramakrishna R, Fontaine D, Sedat J, Lonjon M, Paquis P. Intraventricular fibrinolysis for severe aneurysmal intraventricular hemorrhage: a randomized controlled trial and meta-analysis. Neurosurg Rev. 2013 Oct;36(4):523-30; discussion 530-1. doi: 10.1007/s10143-013-0469-7. Epub 2013 May 2. PMID 23636409